CLINICAL TRIAL: NCT03530163
Title: Breathing Training to Improve Human Performance at High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-0464
Record Dates: First submitted 2018-05-03; First posted 2018-05-21 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Mountain Sickness Acute
Keywords: Exercise; Aerobic; Cognitive Function
MeSH Terms: conditions — Altitude Sickness; Motor Activity | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked from knowing whether they are performing the Respiratory Muscle Training or sham training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory Muscle Training (Experimental)
  Interventions: Device: Respiratory Muscle Training
- Sham Breathing Training (Sham Comparator)
  Interventions: Device: Sham Breathing Training

INTERVENTIONS:
Device: Respiratory Muscle Training — Subjects will breathe through a custom isocapnic Respiratory Muscle Training method developed in-house. The initial breathing frequency will be 30 breaths per minute. Subsequent sessions will begin with 20 minutes of breathing at the highest rate attained on the previous training day. During the last 10 minutes of each session, breathing rate will increase by 1-2 breaths/min.
  Arms: Respiratory Muscle Training
Device: Sham Breathing Training — Each subject in the sham group will be prompted to hold his breath for 10 seconds every 30 seconds (two times each minute) while breathing on a circuit visibly identical to that used in Respiratory Muscle Training. The subject will breathe ambient air normally after each breath hold. Each sham session will last 30 minutes total.
  Arms: Sham Breathing Training

SUMMARY:
Individuals traveling to altitudes above 8,000 feet may suffer from impaired exercise and cognitive performance, and acute mountain sickness (AMS). Decreased barometric pressure, which leads to low blood oxygen levels, is the primary cause of these disorders. Symptoms of AMS are characterized by headache, nausea, vomiting, dizziness, fatigue, and difficulty sleeping. The goal of this research is to identify whether Respiratory Muscle Training will improve physical and cognitive performance, and reduce the symptoms of AMS, at simulated high altitude.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Men, ages 18-45 who are able to achieve at least 3.5 watts/kg of body weight during the peak oxygen uptake test

Exclusion Criteria:

* Less than 18 years old
* Greater than 45 years old
* Have a body mass index greater than or equal to 30
* Have been recent smokers (tobacco or e-cigarettes)
* Current recreational or medical marijuana users
* Currently taking any medication (over-the-counter or prescription) or herbal supplements
* Participants who are unable to tolerate drinking only two, 6-ounce caffeinated beverages per day of the study
* Participants who are legally blind
* Participants who have been to altitudes above Denver (1609m or 5280ft), including air travel, in the 3 weeks prior to the start of the study or with plans to do so during the study
* Participants who have suffered a significant head injury, have anemia or sickle cell trait or disease, have active peptic ulcer disease, diabetes, hypertension, heart disease, HIV/AIDS, glaucoma, kidney disease, liver disease/cirrhosis, adrenal gland failure, hyponatremia/hypokalemia, tuberculosis
* Participants who have a current herpes infection or any other current type of viral or bacterial infection
* Participants with seizure disorders or history of migraines

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in exercise performance during acute simulated high-altitude exposure as measured by a peak oxygen uptake test and time to complete a 720kJ (40km) time trial on a Velotron cycle ergometer. | Baseline and during acute simulated high-altitude exposure. (2 days, 12 hours per day)
  Determine whether Respiratory Muscle Training performed 3x a week for 30 minutes per session is effective in improving exercise performance during acute simulated high-altitude exposure.
Change in cognitive function during acute simulated high-altitude exposure as measured by the DANA cognitive test battery. | Baseline and during acute simulated high-altitude exposure. (2 days, 12 hours per day)
  Determine whether Respiratory Muscle Training performed 3x a week for 30 minutes per session improves cognitive function during simulated high-altitude exposure.
Change in incidence and severity of acute mountain sickness during acute simulated high-altitude exposure as determined by the Lake Louise Questionnaire (a diagnostic survey of acute mountain sickness). | Baseline and during acute simulated high-altitude exposure. (2 days, 12 hours per day)
  Determine whether Respiratory Muscle Training performed 3x a week for 30 minutes per session is effective in reducing incidence and severity of AMS during acute simulated high-altitude exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Roach, PhD, Principal Investigator — Director, Altitude Research Center
Locations (1):
- Altitude Research Center, Aurora, Colorado, United States